CLINICAL TRIAL: NCT00437697
Title: Thromboprophylaxis in Critically Ill Patients: a Prospective, Randomized Study Comparing Anti-Xa Activities Following Subcutaneous Administration of 5000 IU and 7500 IU Dalteparin
Brief Title: Thromboprophylaxis in Critically Ill Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 008/2003
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Venous Thromboembolism
Keywords: dalteparin, critically ill, thromboprophylaxis
MeSH Terms: conditions — Venous Thromboembolism; Critical Illness | interventions — Dalteparin

INTERVENTIONS:
Drug: dalteparin

SUMMARY:
Intensive care patients are at high risk to develop deep venous thrombosis and pulmonary embolism. Despite anticoagulation with heparin 7% of ICU patients suffer from this serious complication. Optimal regimens for prevention of VTE have been established in medical patients only and are not known for ICU patients.

It was therefore the aim of this study to compare the bioavailability of a low molecular weight heparin in ICU patients and in medical patients. Furthermore, we looked wether a 50% dose increase resulted in better bioavailability of this drug.

DETAILED DESCRIPTION:
Background: The optimal dose regimen of low molecular weight heparins (LMWH) for thromboprophylaxis in critically ill patients is unknown.

Objectives: We performed a prospective, randomized study to determine anti-Xa activities following subcutaneous administration of 5000 IU or 7500 IU dalteparin for thromboprophylaxis in ICU patients compared with medical patients receiving the standard dose of 5000 IU.

Patients and Methods: Twenty-five ICU patients received 7500 IU (group 1) and 29 ICU patients received 5000 IU dalteparin subcutaneously (group 2) for thromboprophylaxis. Twenty-nine medical patients receiving 5000 IU dalteparin served as control group (group 3).

ELIGIBILITY:
Inclusion Criteria:

* Requirement for prophylactic anticoagulation, patient age ³19 years, creatinine clearance within normal range, prothrombin time >30% and thrombocyte counts >100 G/l.

Exclusion Criteria:

* Estimated time of admission less than 24 hours, full anticoagulation, renal failure, history of heparin-induced thrombocytopenia, hereditary or acquired coagulation disorders.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-04; Study Completion 2005-04

PRIMARY OUTCOMES:
Area under the curve of measured anti-Xa activities between baseline and 12 hours (AUC-anti-Xa0-12).

SECONDARY OUTCOMES:
Peak anti-Xa activities at any time (C-max anti-Xa)
Time of peak anti-Xa-activities (t-max anti-Xa).

CONTACTS AND LOCATIONS:
Overall Officials: Ute Priglinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria